CLINICAL TRIAL: NCT04550728
Title: Assessment Followed by Home-based Hybrid Robot + FES Rehabilitation Post-stroke
Brief Title: Hybrid Robot+FES Stroke Rehabilitation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00089895
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: stroke; functional electrical stimulation; robot training
MeSH Terms: conditions — Stroke | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FES+robot (Experimental): Participants in this group will have FES during ankle robot training
  Interventions: Combination Product: Ankle robot training and functional electrical stimulation(FES) group
- Robot (Active Comparator): Participants in this group will have ankle robot training only
  Interventions: Combination Product: Ankle robot training group

INTERVENTIONS:
Combination Product: Ankle robot training group — Patients will be seated with the paretic foot strapped to the footplate the knee at full extension. The operator will set up and measure (using the robot) ankle passive DF and PF ROM limits. The robot training will include passive stretching, robot interactive game-based training, and cool-down stretching.
  Arms: Robot
Combination Product: Ankle robot training and functional electrical stimulation(FES) group — Patients will use the ankle robot device as the ankle training group. Also, water-based FES electrodes positioned inside a soft garment will be secured over the DF and PF muscles by wrapping the garment around the leg just below the knee joint. Stimulation intensity will be increased to maximal tolerance of each participant. Electrically induced contraction timing will be triggered by the ankle robot in synchrony with the ankle dorsi and plantar flexion movements.
  Arms: FES+robot

SUMMARY:
The investigators have developed a novel robot-guided stretching under intelligent control and combine it with active movement training, which helped increase joint ROM, reduce spasticity and joint stiffness, increase muscle force output, and improve locomotion. However, for stroke survivors with sensorimotor impairment, their peripheral muscle may not sufficiently be recruited. Functional electrical stimulation (FES), has been shown its advantage to activate the peripheral muscles for people with neurological conditions. The investigators thus make a hybrid robot-FES rehabilitation system, combining the advantage of robot and FES technologies for stroke motor recovery. The investigators further would like to translate the technologies from lab to home-based training. Thus, the investigators will conduct a randomized, controlled, primarily home-based clinical trial using an ankle robot alone or combined with functional electrical stimulation (FES) to treat sensorimotor and locomotion impairments post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85;
* Able to ambulate at least 10 meters without human assistance, with or without an assistive device
* ≥ 6 months post stroke;
* having a caregiver to assist in training at home.

Exclusion Criteria:

* having expressive and receptive aphasia;
* an inability to follow multi-step commands;
* enrolled in another lower limb rehabilitation program;
* having severe pain in the paralyzed lower-limb;
* >30º ankle plantar flexion contracture;
* Having implanted electronic device such as a pacemaker, spinal cord, or deep brain stimulator because FES may potentially interfere with their functions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Lower Extremity | Baseline
  The assessment is a measure of lower extremity (LE) motor and sensory impairments post-stroke.
Fugl-Meyer Lower Extremity | 6 weeks
  The assessment is a measure of lower extremity (LE) motor and sensory impairments post-stroke.
Fugl-Meyer Lower Extremity | 12 weeks
  The assessment is a measure of lower extremity (LE) motor and sensory impairments post-stroke.
Dorsiflexion active range of motion | Baseline
  Joint ankle active range of motion measured by ankle robot.
Dorsiflexion active range of motion | 6 weeks
  Joint ankle active range of motion measured by ankle robot.
Dorsiflexion active range of motion | 12 weeks
  Joint ankle active range of motion measured by ankle robot.
6 minutes walking test | Baseline
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
6 minutes walking test | 6 weeks
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
6 minutes walking test | 12 weeks
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Medical thickness of medial gastrocnemius muscle and tibial anterior muscle | Baseline
  B-model ultrasound will be used to scan the muscle thickness, and the image will be further proceeded to measure the muscle thickness with unit in centimetres.
Medical thickness of medial gastrocnemius muscle and tibial anterior muscle | 6 week
  B-model ultrasound will be used to scan the muscle thickness, and the image will be further proceeded to measure the muscle thickness with unit in centimetres.
Medical thickness of medial gastrocnemius muscle and tibial anterior muscle | 12 week
  B-model ultrasound will be used to scan the muscle thickness, and the image will be further proceeded to measure the muscle thickness with unit in centimetres.
Muscle fiber pennation angle of medial gastrocnemius muscle and tibial anterior muscle | Baseline
  B-model ultrasound will be used to scan the muscle and the image will be further proceeded to measure the muscle fiber pennation angle with unit in degree.
Muscle fiber pennation angle of medial gastrocnemius muscle and tibial anterior muscle | 6 week
  B-model ultrasound will be used to scan the muscle and the image will be further proceeded to measure the muscle fiber pennation angle with unit in degree.
Muscle fiber pennation angle of medial gastrocnemius muscle and tibial anterior muscle | 12 week
  B-model ultrasound will be used to assess the muscle thickness, muscle fiber pennation angle. Elasticity will be measured using ultrasound elastography.

SECONDARY OUTCOMES:
Timed up-to-go | Baseline
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Timed up-to-go | 6 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Timed up-to-go | 12 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Stroke Rehabilitation Assessment of Movement (STREAM) | baseline
  Stroke Rehabilitation Assessment of Movement Measure (STREAM) provides therapists with a quantitative measurement of motor functioning and basic mobility deficits among patients who had a stroke through the performance of 30 voluntary motor tasks of the upper extremities (UE) and lower extremities (LE).
Stroke Rehabilitation Assessment of Movement (STREAM) | 6 weeks
  Stroke Rehabilitation Assessment of Movement Measure (STREAM) provides therapists with a quantitative measurement of motor functioning and basic mobility deficits among patients who had a stroke through the performance of 30 voluntary motor tasks of the upper extremities (UE) and lower extremities (LE).
Stroke Rehabilitation Assessment of Movement (STREAM) | 12 weeks
  Stroke Rehabilitation Assessment of Movement Measure (STREAM) provides therapists with a quantitative measurement of motor functioning and basic mobility deficits among patients who had a stroke through the performance of 30 voluntary motor tasks of the upper extremities (UE) and lower extremities (LE).
Brief Balance Evaluation Systems Test(Brief-BESTest) | baseline
  The Brief BESTest is a clinical balance assessment tool. It is an abbreviated version of Balance Evaluation Systems Test (BESTest), designed to assess 6 different aspects contributing to postural control in standing and walking.
Brief Balance Evaluation Systems Test(Brief-BESTest) | 6 weeks
  The Brief BESTest is a clinical balance assessment tool. It is an abbreviated version of Balance Evaluation Systems Test (BESTest), designed to assess 6 different aspects contributing to postural control in standing and walking.
Brief Balance Evaluation Systems Test(Brief-BESTest) | 12 weeks
  The Brief BESTest is a clinical balance assessment tool. It is an abbreviated version of Balance Evaluation Systems Test (BESTest), designed to assess 6 different aspects contributing to postural control in standing and walking.
Modified Ashworth Scale (MAS) | baseline
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
Modified Ashworth Scale (MAS) | 6 weeks
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
Modified Ashworth Scale (MAS) | 12 weeks
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
10-meter walk test (10MWT) | baseline
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
10-meter walk test (10MWT) | 6 weeks
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
10-meter walk test (10MWT) | 12 weeks
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Stiffness of medial gastrocnemius muscle and tibial anterior muscle. | Baseline
  Supersonic shear wave elastography will be used to estimate the shear wave speed(m/s) of the muscles.
Stiffness of medial gastrocnemius muscle and tibial anterior muscle. | 6 weeks
  Supersonic shear wave elastography will be used to estimate the shear wave speed(m/s) of the muscles.
Stiffness of medial gastrocnemius muscle and tibial anterior muscle. | 12 weeks
  Supersonic shear wave elastography will be used to estimate the shear wave speed(m/s) of the muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang LQ, Chung SG, Bai Z, Xu D, van Rey EM, Rogers MW, Johnson ME, Roth EJ. Intelligent stretching of ankle joints with contracture/spasticity. IEEE Trans Neural Syst Rehabil Eng. 2002 Sep;10(3):149-57. doi: 10.1109/TNSRE.2002.802857. PMID 12503779
- [Background] Selles RW, Li X, Lin F, Chung SG, Roth EJ, Zhang LQ. Feedback-controlled and programmed stretching of the ankle plantarflexors and dorsiflexors in stroke: effects of a 4-week intervention program. Arch Phys Med Rehabil. 2005 Dec;86(12):2330-6. doi: 10.1016/j.apmr.2005.07.305. PMID 16344031
- [Background] Ren Y, Wu YN, Yang CY, Xu T, Harvey RL, Zhang LQ. Developing a Wearable Ankle Rehabilitation Robotic Device for in-Bed Acute Stroke Rehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2017 Jun;25(6):589-596. doi: 10.1109/TNSRE.2016.2584003. Epub 2016 Jun 22. PMID 27337720
- [Background] Embrey DG, Holtz SL, Alon G, Brandsma BA, McCoy SW. Functional electrical stimulation to dorsiflexors and plantar flexors during gait to improve walking in adults with chronic hemiplegia. Arch Phys Med Rehabil. 2010 May;91(5):687-96. doi: 10.1016/j.apmr.2009.12.024. PMID 20434604